CLINICAL TRIAL: NCT03944330
Title: A Clinic Trail on Nutrition Support Therapy of Patients With Liver Failure
Brief Title: A Study on Nutrition Support Therapy of Patients With Liver Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qin Ning, Director and Chair of Department of Infectious Diseases, Tongji Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Nstlf
Record Dates: First submitted 2019-03-14; First posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a treatment group (Active Comparator): All study participants were provided with a standard hospital diet that provided B25-30 kcal/kg/day
  Interventions: Dietary Supplement: standard hospital diet
- control group (No Intervention): All study participants were not intervened with diet

INTERVENTIONS:
Dietary Supplement: standard hospital diet — patients were provided standard hospital diet that provided 25-30 kcal/kg/day
  Arms: a treatment group

SUMMARY:
This study is a Clinical trial to assess the efficacy of nutrition support therapy of patients with liver failure. Patients were randomized to one of 2 groups to receive different nutrition and energy support treatment.

DETAILED DESCRIPTION:
Patients with liver failure (defined by APASL) induced by any precipitating factors were randomized to two groups; a treatment group and a control group. Participants in treatment group were provided with a standard hospital diet that provided 25-30 kcal/kg/day . Patients in control group receive diet guide

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients from 18 to 65 years of age;
2. Patient inclusion criteria: jaundice (serum total bilirubin ≥5 mg/dl) and coagulopathy (INR ≥ 1.5 or prothrombin activity ≥ 40 %), accompanied by ascites and/or encephalopathy within 4 weeks.

Exclusion Criteria:

1. Surgery with in 4 weeks
2. three degree hepatoencephalopathy
3. malignant tumors
4. cardiac failure or respiratory failure
5. liver transplantation within observing period -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-10 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Mortality at 30 day | 4 weeks
  The percentage of death of liver failure patients at 4 weeks

SECONDARY OUTCOMES:
liver transplant-free survival | 3month
  survival rate on 4 weeks and 3 month
Laboratory variables on serum biochemistry markers | 3month
  Laboratory variables on serum lever of glutamic-pyruvic transaminase/glutamic oxalacetic transaminase/total bilirubin/ cholinesterase will be combined to report liver function
Laboratory variables on fasting blood sugar | 3month
  Laboratory variables on serum lever of fasting blood sugar

IPD SHARING:
Plan to Share IPD: No